CLINICAL TRIAL: NCT06335056
Title: Dissemination of an Adolescent Obesity Prevention Intervention to Louisiana Schools
Acronym: ProudMe
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University and A&M College (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Pennington Biomedical Research Center (Other); Texas A&M University (Other); University of Nevada, Las Vegas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRBAM-21-0702; 1R15HD108765-01A1 (NIH)
Record Dates: First submitted 2024-02-26; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Treatment (ProudMe); Waitlist Control

STUDY DESIGN:
Intervention Model Description: In this 12-week long intervention project, 480 adolescent participants are randomized, at the school level, to 2 arms - ProudMe or waitlist control conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ProudMe (Experimental): The ProudMe condition involves three key components: (a) artificial intelligence (AI)-assisted behavior management system (i.e., ProudMe Tech), (b) ProudMe physical/health education (PE) and lunchroom reform (ProudMe Cafeteria), (c) customized implementation training (ProudMe Training).
  Interventions: Behavioral: ProudMe
- Waitlist Control (Active Comparator): The waitlist control involves (a) regular physical/health education and lunchroom, (b) professional development training on the importance of quality physical/health education, health eating and foot environment. It does not involve AI-assisted behavior management system.
  Interventions: Behavioral: Waitlist Control

INTERVENTIONS:
Behavioral: ProudMe — ProudMe Tech: Regular human/computer interaction (3-5 times per week) to engage in SMART goal-setting, behavior monitoring, and self-reflection as assisted by AI-enabled feedback.
  ProudMe Physical Education [PE]: 12 lessons to acquire knowledge, skill, and dispositions to improve physical activity, diet, screen-based sedentary behaviors.
  ProudMe Cafeteria: Purposely enabling policy and environmental changes in school cafeteria (recognize areas of strengths and weaknesses; set goals and action plans; make changes to improve scores assessed by the Smarter Lunchroom Scorecard).
  ProudMe Training: 4-hour implementation training + regular check-in and support (via motivational interviewing techniques)
  Arms: ProudMe
Behavioral: Waitlist Control — The waitlist control involves (a) regular physical/health education and lunchroom, (b) professional development training on the overall importance of quality physical/health education, health eating and foot environment. It does not involve AI-assisted behavior management system.
  Arms: Waitlist Control

SUMMARY:
This project aims to test the effectiveness and implementation of an adolescent obesity prevention intervention called ProudMe. The study recruits 480 adolescents from 12 middle schools (cluster-randomized to 6 ProudMe schools vs 6 wait-list control schools) and expect to observe improvements of obesity-prevention behaviors and weight status in the ProudMe group compared to the control. The investigators also collect mixed-methods data from 24 school implementers at the 6 ProudMe schools and expect to observe appropriate levels of adaptation, fidelity, reach, penetration, and sustainability, with manageable time and financial cost.

DETAILED DESCRIPTION:
The Louisiana-based, 12-week, multi-level, multi-component, ecological intervention is called Preventing Obesity Using Digital-assisted Movement and Eating (ProudMe). Guided by robust theories and prior work, this project involves multiple trained student researchers to address two specific aims.

Aim 1: to test the effectiveness of the ProudMe intervention in Louisiana middle schools. Informed by power analysis (80% statistical power), the study recruits 480 adolescents from 12 middle schools (cluster-randomized to 6 ProudMe schools vs 6 wait-list control schools). Quantitative data on obesity-prevention behaviors (i.e., physical activity, screen-based sedentary behavior, diet behaviors) and weight status (i.e., body mass index z score, waist circumference) are collected from all adolescent participants using validated instruments and procedures. The investigators hypothesize the multi-level modeling analyses to show improvements of obesity-prevention behaviors and weight status in the ProudMe group compared to a waist-list control, after controlling for sociodemographic factors at multiple ecological levels.

Aim 2: to test the implementation outcomes of the ProudMe intervention in Louisiana middle schools. The investigators collect mixed-methods data from 24 school implementers (i.e., teachers, administrators, and staff), 96 adolescents, and 96 parents at the 6 ProudMe schools, to capture adaptation and implementation indicators. The investigators evaluate the adaptations made across three phases (early, mid, late) of the implementation (i.e., what, at what level, when, how, why, by whom, and impact to intervention). In addition, the investigators assess reach, fidelity, penetration, sustainability, and cost of the implementation across early, mid, and late phases of the implementation. The investigators expect the ProudMe schools to show appropriate levels of adaptation, fidelity, reach, penetration, and sustainability, with manageable time and financial cost.

Building on previously funded work (e.g., R21HD090513, PI: Dr. Chen), this project is led by a strong, collaborative, transdisciplinary team with experts from kinesiology, developmental psychology, nutrition, childhood obesity, computer science, statistics, and implementation science. The project significantly strengthens the research environment of the Louisiana State University (LSU) - a primarily undergraduate student serving institution under-funded by the NIH. The project creates unique opportunities that are otherwise unavailable for LSU students who aspire to seek advanced education or careers in biomedical and health fields.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in 6th, 7th, or 8th grades in participating schools.
* Students with parental consent and child assent.

Exclusion Criteria:

* Students enrolled in grades other than 6th, 7th, or 8th grades
* Students in non-participating schools.
* Students without parental consent and child assent.
* Students without adequate readiness for physical activity.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — All genders are eligible to participate in the study.
Enrollment: 480 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Physical activity: NHANES physical activity recall question, Leisure-Time Exercise Questionnaire, ActiGraph accelerometers | 12 weeks
  Self-reported screen time
Screen time | 12 weeks
  a screen time questionnaire
Food environment | 12 weeks
  Parent-reported Food Frequency Questionnaire

SECONDARY OUTCOMES:
Body mass index z score | 12 weeks
  Body mass index (BMI) z scores and BMI scores are converted by weight and height. Body weight is measured to the nearest 0.1kg with a calibrated Seca Model 770 scale. Raw BMI score is calculated from height and body weight as follows: BMI (kg/m2) = Body weight (kg) / Height (m)2. BMI-z score is calculated to examine how many standard deviations adolescents' BMI is above or below the average BMI value for their age group and gender.
Waist circumference | 12 weeks
  Waist circumference at the umbilicus is assessed to the nearest 0.5cm using a constant tension tape.

OTHER OUTCOMES:
Activity self-efficacy | 12 weeks
  An individual-level covariate. Activity self-efficacy refers to adolescents' belief in their capability to participate in physical activity despite barriers. Adolescent participants will complete an 8-item activity self-efficacy measure, to assess activity self-efficacy during free time on most days overall, despite barriers (screen time, weather, location, schedule, social support).
Self-monitoring | 3-5 times per week over 12 weeks
  An individual-level covariate. Adolescent participants set up daily goals for physical activity, screen time, dietary behaviors, and sleep; track their behavior efforts, and evaluate goal attainment on the ProudMe Tech system.
Social support | 12 weeks
  An interpersonal-level covariate. To assess the sources and types of social support.
School Wellness Policy | 12 weeks
  The Wellness School Assessment Tool 3.0 (WellSAT 3.0) to assess environmental/policy changes in schools (pre to post tests).
Cafeteria Nutrition | 12 weeks
  School Cafeteria Nutrition Assessment (SCNA) to evaluate the lunch menus and observe foods offered in the cafeteria (monthly).

CONTACTS AND LOCATIONS:
Locations (1):
- LSU Pedagogical Kinesiology Lab, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No